CLINICAL TRIAL: NCT04386681
Title: Re-entry Continuum for Brain Injury
Acronym: RCBI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rehabilitation Hospital of Indiana (Other)
Responsible Party: Principal Investigator, Devan Parrott, Director of the Research Training and Outcome Center, Rehabilitation Hospital of Indiana
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1909189045
Record Dates: First submitted 2020-04-27; First posted 2020-05-13 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Traumatic Brain Injury; Recidivism
Keywords: Offenders
MeSH Terms: conditions — Brain Injuries, Traumatic; Recidivism

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RCBI (Experimental): Receiving RCBI intervention, including BICS, ICAN, and RF.
  Interventions: Behavioral: Reentry Continuum for Brain Injury (RCBI)
- Treatment as usual- Control group (No Intervention): Not receiving the RCBI intervention

INTERVENTIONS:
Behavioral: Reentry Continuum for Brain Injury (RCBI) — Pre-Release RCBI Treatment Procedures (BICS and ICAN). BICS: consists of 12 weekly two- hour sessions. Sessions focus on brain injury education, coping skills for the various symptoms of brain injury, depression management, stress management, and self- advocacy.
  ICAN: delivered once a week for 6 weeks for 2 hours per session. ICAN primarily focuses on poor perspective-taking and inability to make social inferences about others' behaviors that are related to negative attributions, and employs role playing exercises and a novel perspective-positioning technique to elicit affective and cognitive empathy to alter negative attributions and reduce anger.
  Post-Release RCBI Resource Facilitation. Working with their resource facilitator, alongside their corrections case manager, to work on brain injury specific reentry planning, resource, and needs identification.
  Arms: RCBI

SUMMARY:
The overall research objectives of the proposed project are to decrease the rate of recidivism, defined as returning to incarceration within three years of release, as well as reduce the number of violent offenses, through the successful implementation of a continuum of services that addresses the unique needs of the TBI population. RHI, in partnership with PCF and IU, will work together to accomplish these goals. To meet study objectives, this randomized controlled trial (RCT) will enroll 102 individuals with TBI who will be randomized into the Reentry Continuum for Brain Injury (RCBI) intervention or a TAU-CG. Participants will be screened for TBI eight months prior to release from PCF. Upon consenting to participate, all subjects will be evaluated before, during, and after the intervention and recidivism data will be collected through IDOC's Data Analysis and Technology Department.

DETAILED DESCRIPTION:
Specific aims of the current proposal are as follows:

Aim 1. To examine differences in recidivism [return to incarceration within 3 years] in participant offenders with TBI who are reentering the community and are either randomized to RCBI or TAU-CG.

Hypothesis 1 (H1): Participants in the RCBI group will demonstrate a lower proportion of recidivating participants than the TAU-CG one year, two years, and three years post release.

Aim 2. To examine differences in violent offenses [number of pre-release violent behavioral infractions; number of post-release felonies committed and their classifications] in participant offenders with TBI who are reentering the community and are either randomized to RCBI or TAU-CG during 3 months pre-release, and one, two, and three years post-release.

Hypothesis 2A (H2A): Participants in the RCBI group will demonstrate lower rates of in-prison violent behavioral infractions between enrollment and release than participants in the control group.

Hypothesis 2B (H2B): Participants in the RCBI will commit fewer and less serious level felonies post-release than participants in the TAU-CG 1, 2, and 3 years post-release demonstrated by a lower proportion of RCBI offenders committing violent crimes than TAU-CG.

Aim 3. Examine group differences in coping [Brain Injury Coping Skills Questionnaire], aggression [Buss Perry Aggression Questionnaire], community integration [Participation Assessment with Recombined Tools-Objective], and number of basic needs unmet [Survey of Unmet Needs and Services] at time of release and 1-year post-release as well as employment [Employment acquisition and sustainability] 1, 2, and 3 years post-release.

Hypothesis 3A (H3A): Participants in the treatment group will show better scores on measures of coping and aggression compared to controls at time of release.

Hypothesis 3B (H3B): The RCBI group will show a higher proportion of participants obtaining employment compared to the TAU-CG as well as higher employment durations (total months showing employment data) one year, two years, and three years post release and better community integration one-year post release.

Hypothesis 3C (H3C): Participants in the treatment group will show lower rates of unmet needs compared to the control group one-year post release.

Aim 4 (Exploratory). Identify which factors predict recidivism in the TBI population and investigate their relationship with a validated measure of recidivism risk [Level of Service Inventory-Revised7].

Hypothesis 4 (H4): While it is hypothesized that group assignment (RCBI vs. TAU-CG) in combination with criminality risk and select demographic, injury, and/or social variables will contribute significantly to a model predicting three-year recidivism outcome, a specific model is not hypothesized and detection of specific contributing variables will be exploratory.

ELIGIBILITY:
Inclusion Criteria:

* History of moderate to severe TBI
* Ages 18 and older
* Offenders currently serving their sentence at PCF in Greencastle, Indiana
* Approximately twelve or less months remaining in their sentence, but no fewer than 5 months remaining in sentence.

Exclusion Criteria:

* In restricted housing (e.g., solitary confinement)
* Inability to comprehend the study
* Individuals requiring a legally authorized representative (LAR)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in Brain Injury Coping Skills Questionnaire (BICS-Q) | within 2 weeks, 3 months
  Designed to measure self-efficacy related to brain injury. BICS-Q was designed based on Bandura's Guide for developing self-efficacy scales. Participants rate 20 items using a 5-point Likert-scale resulting in a total score. BICS-Q has shown significant change across BICS participants in multiple studies. Participants rate each statement from 0 (Not at all) to 4 (Extremely). Higher scores suggest greater self-efficacy.
Change in Aggression Questionnaire (AQ) | within 2 weeks, 3 months
  A standardized measure comprised of 34 statements to assess anger, hostile thoughts, and physical and verbal aggression.10 Participants rate statements using a 5-point scale (1 - Extremely uncharacteristic of me to 5 - Extremely characteristic of me). Raw and scaled scores (adjusted by age and gender) are provided for aggression subcomponents and total aggression. Total aggression will be used for our analyses. The AQ is a widely used measure, including for TBI studies.11 It has good test-retest reliability (.72-.80), and good internal consistency (.76-.94). Higher scores suggest higher aggression tendencies
Change in Attributions of Intent Hostility Questionnaire (AIHQ) | within 2 weeks, 3 months
  This consists of 5 written vignettes describing ambiguous actions/ situations (unclear intent behind actions). After participants read each vignette and imagine the scenario happening to her or him, they are asked five questions: 1) why the other person (or persons) acted that way toward you (open-ended response later rated by an independent rater; score indicates ''hostility bias''); 2) Whether the other person (or persons) performed the action on purpose (1 ''definitely no'' to 6 ''definitely yes'') using a Likert Scale (Intent score); 3) how angry it would make them feel (1 ''not at all angry'' to 5 ''very angry'') using a Likert scale (anger score); 4) how much they would blame the other person (or persons) (1 ''not at all'' to 5 ''very much'') using a Likert scale (blame score); and 5) how she or he would respond to the situation, (open-ended response).
Change in Participation Assessment with Combined Tools - Objective (PART-O) | 3 months, 1 year
  This is a 17-item measure developed and validated by the NIDILRR-sponsored TBI Model Systems13 to evaluate participation in the community with three domains: Productivity, Social Relations, and Out and About. Each item is scored on a 0 to 5 scale. Total PART-O scores will be used for our analyses.
Change in Survey of Unmet Needs and Services Utilized (SUNSU) | 3 months, 1 year
  This measure is designed to assess both the usage of and desire for services unique to brain injury. The SUNSU includes a comprehensive list of 27 service needs and results in two scores: the number of met needs and the number of unmet needs. The measure shows good internal consistency as well as validity when compared to other needs assessments in the brain injury population. Participants decide if they : currently want help for the need, currently receiving help for the need, or it is not a need at all.
Change in Recidivism | 1 year after release, 2 years after release, 3 years after release
  This is defined as return to incarceration within three years of release and is the primary outcome to be collected through the IDOC Research and Technology Division for all participants at three time points: one, two, and three years after release.
Change in Behavioral Infractions | 3 months
  This is collected from PCF directly for each participant at time of release. The number and type of infractions will be counted between study enrollment and release.
Change in Employment | Prior to release, 1 year after release, 2 years after release, and 3 years after release
  This includes acquisition and sustainability (i.e., duration of employment) data will be collected through the IDOC Research and Technology Division for all offenders at three time points: one year, two years, and three years after release from IDOC.
Change in Violent Rearrests | 1 year after release, 2 years after release, 3 years after release
  This is collected for each participant through the IDOC Data Analysis and Technology Department for all offenders at three time points: one year, two years, and three years after release from IDOC. Offenses are coded between 1 and 6 with 1 being the highest level of violence and 6 being the lowest level/non-violent. Type of offense in criminal history (violent vs. nonviolent) will also be collected as a covariate.

SECONDARY OUTCOMES:
Level of Service Inventory - Revised (LSI-R) | within 2 weeks
  This is a 54-item scale designed to measure criminal risk with ten subscales of criminogenic factors including Criminal History, Education/Employment, Financial, Family Marital, Accommodation, Leisure/Recreation, Companions, Alcohol/Drug Problems, Emotional/Personal, and Attitudes/Orientation. The items are scored utilizing a dichotomous rating system of 0 = absent and 1 = present with final scores ranging from 0 to 54. The LSI-R has been studied extensively and is considered one of the most used risk assessments in the offender population.15 Inter-rater reliability coefficients range from .80 to .96 with studies of validity showing that higher LSI-R scores have been associated with recidivism (short- and long-term), adjustment, and institutional misconduct. Higher scores suggest greater likelihood of recidivism, criminality, substance use, etc.
Change in Behavioral Rating Inventory of Executive Function-Adult Version (BRIEF-A) | within 2 weeks, 3 months, 1 year
  This is a standardized measure published by Psychological Assessment Resources (PAR) designed to measure self-regulation in adults. The BRIEF-A consists of 75 items, takes 10 to 15 minutes to administer and generates nine subscales: Inhibit, Self-Monitor, Plan/Organize, Shift, Initiate, Task Monitor, Emotional Control, Working Memory, and Organization of Materials. Participants rate each item as 0 = Never, 1 = Sometimes, 2 = Often.

CONTACTS AND LOCATIONS:
Overall Officials: Devan Parrott, PhD, Principal Investigator — Indiana University
Locations (1):
- Putnamville Correctional Facility, Greencastle, Indiana, United States

IPD SHARING:
Plan to Share IPD: No